CLINICAL TRIAL: NCT02996318
Title: Treatment of Coronary In-Stent Restenosis by a Sirolimus (Rapamycin) Coated Balloon or a Paclitaxel Coated Balloon
Acronym: FIMLIMUSDCB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InnoRa GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SI01
Record Dates: First submitted 2016-12-09; First posted 2016-12-19 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: DES In-stent Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus coated Balloon (Experimental): treatment of coronary DES-ISR with a sirolimus coated balloon
  Interventions: Device: Sirolimus coated balloon
- Paclitaxel coated balloon (SeQuent Please) (Active Comparator): treatment of coronary DES-ISR with a paclitaxel coated balloon
  Interventions: Device: Paclitaxel coated balloon (SeQuent Please)

INTERVENTIONS:
Device: Paclitaxel coated balloon (SeQuent Please) — Paclitaxel coated balloon (SeQuent Please)
  Arms: Paclitaxel coated balloon (SeQuent Please)
Device: Sirolimus coated balloon — Sirolimus coated balloon
  Arms: Sirolimus coated Balloon

SUMMARY:
The aim of the study is to investigate the non-inferiority of the new sirolimus-coated balloon catheters in comparison to the paclitaxel-coated SQP with regard to acute tolerance, safety and efficacy in coronary DES in-stent restenosis.

DETAILED DESCRIPTION:
The aim of the study is to investigate the non-inferiority of the new sirolimus-coated balloon catheters in comparison to the paclitaxel-coated SQP with regard to acute tolerance, safety and efficacy in coronary DES in-stent restenosis.

Patient population will consist of male and female adults suffering from coronary drug-eluting stent (DES) restenosis, which is to be treated by a study balloon according to the inclusion and exclusion criteria as defined below.

In Late lumen loss lesion (difference between the angiographic in-lesion MLD post procedural and at 6 months follow-up) will be evaluated by quantitative coronary angiography (QCA).

The study will be performed as a single-blind, SQP controlled study in 4 - 6 study centers in 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Clinical evidence of stable or unstable angina (acute coronary syndrome) or a positive functional study
* Patients with ≤ 2 primary drug-eluting stent in-stent restenosis (DES-ISR) lesions (≥ 70% diameter stenosis by visual estimation or ≥ 50% and positive functional study) including margin stenosis with max 5mm distance to the stent.

Exclusion Criteria:

* Chronic renal insufficiency with serum creatinine levels > 2.0 mg per deciliter
* Known hypersensitivity or contraindications to aspirin, heparin, clopidogrel, ticlopidine or sirolimus, and sensitivity to contrast media not amenable to premedication
* Concomitant medical illness associated with a life-expectancy of less than two year
* Lesion length (ISR) > 35 mm, vessel diameter < 2.5 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Late lumen loss | 6 months
  Difference between minimal lumen diameter at follow-up coronary angiography and baseline after PCI

SECONDARY OUTCOMES:
Procedural Success | 24 hours
  ≤ 30% final stenosis, TIMI III flow, no flow-limiting dissection at the conclusion of the procedure, and the absence of in-hospital (24 hour after treatment) MACE
MACE (Major adverse cardiac events) | 12 months
  MACE will be defined as the occurrence of cardiac death, target vessel myocardial infarction, or clinically driven target lesion revascularization at 6 months and 12 months.

CONTACTS AND LOCATIONS:
Locations (5):
- Malaysia (5):
  - Queen Elizabeth Hospital II, Kota Kinabalu
  - National Heart Institute, Kuala Lumpur
  - University Malaya, Kuala Lumpur
  - Sarawak Genaral Hospital Heart Centre, Kuching
  - Hospital Pulau Pinang, Pulau Pinang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scheller B, Mangner N, Abdul Kader MASK, Wan Ahmad WA, Jeger R, Wohrle J, Ong TK, Liew HB, Gori T, Mahfoud F, Nuruddin AA, Woitek F, Abidin IZ, Schwenke C, Schnorr B, Mohd Ali R. Combined Analysis of Two Parallel Randomized Trials of Sirolimus-Coated and Paclitaxel-Coated Balloons in Coronary In-Stent Restenosis Lesions. Circ Cardiovasc Interv. 2022 Sep;15(9):e012305. doi: 10.1161/CIRCINTERVENTIONS.122.012305. Epub 2022 Sep 20. PMID 36126132
- [Derived] Ali RM, Abdul Kader MASK, Wan Ahmad WA, Ong TK, Liew HB, Omar AF, Mahmood Zuhdi AS, Nuruddin AA, Schnorr B, Scheller B. Treatment of Coronary Drug-Eluting Stent Restenosis by a Sirolimus- or Paclitaxel-Coated Balloon. JACC Cardiovasc Interv. 2019 Mar 25;12(6):558-566. doi: 10.1016/j.jcin.2018.11.040. PMID 30898253